CLINICAL TRIAL: NCT06889831
Title: Adaptation of a Digital Group-Based Intervention to Reduce Drug Use and Increase Contraceptive Use Among Reproductive-Aged Women Involved in Criminal Justice Systems
Brief Title: WORTH Paths Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fairleigh Dickinson University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Melissa Slavin, Assistant Professor, Fairleigh Dickinson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FDU-K01-2022-MNS; 5K01DA055762-04 (NIH)
Record Dates: First submitted 2025-03-09; First posted 2025-03-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Substance Use Disorder (SUD); Sexual and Reproductive Health; Sexual Risk Behavior
Keywords: substance use disorder
MeSH Terms: conditions — Substance-Related Disorders; Coitus

STUDY DESIGN:
Intervention Model Description: Parallel Assignment - Participants will be randomly assigned to one of two groups:
  * Intervention Group: Receives a digital intervention including facilitated group-based treatment via videoconference and interactive activities to reduce substance use and improve contraceptive use.
  * Control Group: Receives a wellness intervention focusing on stress reduction, physical activity, and general health.
  This is a pilot randomized controlled trial. The study will recruit 50 reproductive-aged women involved in criminal legal systems with substance use disorders and unmet need for contraception who will be randomly assigned to either the intervention (n=25) or the wellness control condition (n=25). Both arms involve facilitated group-based treatment via videoconference.
Masking Description: N/A (No masking in this study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WORTH Paths Digital Intervention Group (Experimental): Participants will receive a culturally tailored program adapted for reproductive-aged women involved in the criminal legal system with substance use disorders and unmet contraceptive needs. The intervention consists of three facilitated group sessions over videoconference with digital interactive activities to support behavior change.
  Key components include:
  * Raising awareness about different contraceptive methods and substance use treatment options
  * Discussing personal motivations for reducing drug use and using contraception
  * Developing skills to identify and manage substance use and reproductive health triggers
  * Digital interactive activities to reinforce learning and skill-building
  * Practicing decision-making tools and goal-setting strategies
  * Addressing barriers related to safety including intimate partner violence
  * Creating a safety plan and strategies for maintaining progress
  * Resources for state and online substance use and sexual/reproductive health services
  Interventions: Behavioral: WORTH Paths Digital Intervention
- WORTH Paths Digital Wellness Group (Active Comparator): Participants in this arm will receive the WORTH Paths Wellness Group, a wellness-focused intervention delivered via three facilitated group sessions over videoconference with digital interactive activities. Sessions cover general health, stress reduction, and navigating health services. Topics include education about substance use and sexual and reproductive health risks, guided meditation and mindfulness training, stress management techniques, and an overview of substance use and reproductive health services. Participants will also receive digital wellness resources, including recorded mindfulness exercises and links to online platforms for health services.
  Interventions: Behavioral: WORTH Paths Wellness Group

INTERVENTIONS:
Behavioral: WORTH Paths Digital Intervention — Participants in this arm will receive the WORTH Paths digital intervention, a culturally tailored program designed for women involved in the criminal legal system with substance use disorders and unmet contraceptive needs. The intervention consists of three facilitated group sessions over videoconference with digital interactive activities to support behavior change.
  Arms: WORTH Paths Digital Intervention Group
Behavioral: WORTH Paths Wellness Group — A wellness-focused intervention consisting of three facilitated group sessions over videoconference with digital interactive activities. Sessions cover general health, stress reduction, and navigating health services, including education about substance use and sexual/reproductive health risks, guided meditation, stress management techniques, and an overview of available health services. Participants also receive digital wellness resources, including recorded mindfulness exercises and links to online health service platforms.
  Arms: WORTH Paths Digital Wellness Group

SUMMARY:
Women in the criminal legal system are more likely to experience substance use disorders and unintended pregnancy than women in the general public. However, they often face barriers to accessing substance use treatment and sexual and reproductive health services.

This study tests the feasibility and acceptability of Women on the Road to Health (WORTH) Promoting Access to Treatment, Health, and Support (Paths), a digital intervention adapted from the evidence-based CDC Best Practice HIV prevention intervention, Women on the Road to Health (WORTH), originally developed at Columbia University School of Social Work. WORTH Paths is designed to help reproductive-aged women in the criminal legal system with substance use disorders and unmet need for contraception reduce drug use and improve contraceptive use.

Participants (N=50) will be randomly assigned to one of two groups:

WORTH Paths Intervention Group - Participants will attend three virtual group sessions with facilitated videoconference sessions and self-paced digital activities focused on reducing drug use and increasing contraceptive use. They will also receive guidance on how to access and navigate health services.

Control Group - Participants will receive a virtual general wellness program that includes education on substance use and sexual and reproductive health but does not include skills-based training related to these topics. The focus will be on general wellness and stress reduction.

Both groups will receive resources for substance use treatment and sexual and reproductive health services.

Researchers will track changes in drug use and contraceptive use over three months. Participants will complete surveys and provide urine samples to confirm changes in drug use.

Primary aims:

Feasibility: Measured by session attendance, treatment completion, dropouts, and reasons for termination.

Acceptability: Measured by participant ease of use, helpfulness, and satisfaction.

Primary behavioral outcomes:

Self-reported drug use confirmed by urine drug tests. Contraceptive use, including initiation and consistent use.

Secondary behavioral outcome:

Linkage to substance use disorder treatment (measured by appointments made and sessions attended).

DETAILED DESCRIPTION:
Many women involved in the criminal legal system experience substance use disorders and unintended pregnancy but face significant barriers to accessing and utilizing substance use treatment and sexual and reproductive health services. These barriers include limited social support, intimate partner violence, and challenges with self-advocacy and decision-making regarding substance use treatment and contraception. The siloed nature of healthcare services also makes it difficult for women to receive integrated care that addresses both substance use and sexual and reproductive health needs.

While some existing programs for women in the criminal legal system focus on HIV prevention through condom use, fewer interventions take a comprehensive approach to sexual and reproductive health by addressing all forms of contraception while also integrating substance use treatment strategies.

This study tests WORTH Paths, a digital intervention designed to reduce drug use and increase contraceptive use. WORTH Paths builds on Women on the Road to Health (WORTH), an evidence-based CDC Best Practice HIV prevention intervention originally developed at the Columbia University School of Social Work. While WORTH has been effective in increasing condom use, this new adaptation expands its focus to a broader range of contraceptive methods and strategies to support women in reducing drug use.

Study Design

This study is a randomized controlled trial (RCT). Participants will be randomly assigned to one of two groups:

1. WORTH Paths Intervention Group

   Participants in this group will receive the WORTH Paths program, a culturally tailored digital intervention designed to help women involved in the criminal legal system reduce substance use and improve contraceptive use. This intervention includes:
   * Three virtual group sessions led by trained facilitators via videoconferencing
   * Culturally relevant digital interactive activities, including animations, videos, and exercises to reinforce key skills
   * Education on a full range of contraceptive methods, including long-acting reversible contraception (LARC), barrier methods, and other effective forms of contraception at reducing unintended pregnancy and sexually transmitted infections
   * Guidance on accessing and navigating substance use treatment and reproductive healthcare services, including how to advocate for their needs within the healthcare system
   * Cognitive-behavioral and motivational interviewing (MI)-based activities to help participants develop personalized strategies for reducing substance use and improving reproductive health behaviors
   * Skill-building for self-regulation and behavioral strategies, including managing drug-related triggers, coping with relationship and environmental stressors, and setting personal health goals
   * Safety planning and decision-making strategies, with a focus on reducing interpersonal risks such as intimate partner violence and reproductive coercion
   * Participants in the intervention group will also receive resources for substance use treatment and sexual and reproductive health services, including referrals to local and online providers for contraception and substance use treatment.
2. Control Group (Wellness Program)

Participants in the control group will receive a general wellness program designed to provide support and education while excluding the behavioral skill-building components of the intervention. This program includes:

* Three virtual group sessions led by trained facilitators via videoconferencing
* Education about challenges in accessing substance use treatment and sexual and reproductive health services among women in the criminal legal system
* Guided mindfulness exercises, including meditation and relaxation techniques
* Stress management strategies, such as breathing exercises and coping mechanisms for managing emotional distress
* General wellness discussions on self-care and maintaining overall well-being
* Referrals and informational resources for substance use treatment and reproductive health services, but no structured training on how to navigate or advocate for care Unlike the intervention group, the control group will not receive training in behavioral change strategies related to substance use or contraceptive use.

Assessments & Data Collection

All participants will complete:

* Baseline assessments and mail-in urine drug tests at enrollment
* Follow-up assessments and mail-in urine drug tests at 3 months
* Participants will report on drug use and contraceptive use through online surveys. Urine samples will biologically verify changes in drug use.

Eligibility Criteria

To participate, individuals must:

* Identify as a woman aged 18-44
* Have had criminal legal system involvement within the past year
* Meet DSM-5 criteria for current illicit substance use disorder as assessed by the Mini International Neuropsychiatric Interview (MINI)
* Have a past 30-day history of unmet need for contraception (not using contraception despite not wanting to become pregnant)
* Live in the New York metropolitan area (New York, New Jersey, or Connecticut)

Exclusion Criteria:

* Unable to give informed consent due to a medical condition or cognitive impairment
* Does not speak, read, or write in English
* Unwilling to follow study procedures Recruitment Methods
* Participants will be recruited through community-based organizations that serve formerly incarcerated women. Recruitment efforts will include:

Flyers and posters at community centers and shelters

* Announcements on community listservs
* Direct referrals from program staff
* Participation is completely voluntary, and participants may withdraw at any time. Privacy will be strictly protected.

Data Collection & Safety Measures The study will use self-reported surveys and urine drug tests to measure changes in substance use.

Surveys will be completed securely online

* Data will be stored in a password-protected, encrypted system to ensure confidentiality
* Trained facilitators will monitor sessions and provide referrals if needed. If a participant experiences distress, they will be connected to counseling and substance use treatment resources.

Potential Benefits

While there is no guaranteed benefit, participants may:

* Gain new knowledge about contraception and reproductive health
* Receive support and strategies for reducing drug use and improving contraceptive use
* Obtain referrals for substance use treatment and sexual/reproductive health services (local and online)
* Improve self-efficacy and decision-making skills

ELIGIBILITY:
Inclusion Criteria:

* Female sex at birth
* Aged 18-44 years
* Past year criminal legal involvement (e.g., incarceration or community supervision)
* Meets criteria for current substance use disorder (SUD) as defined by DSM-5 and assessed by the Mini-International Neuropsychiatric Interview (MINI)
* Meets criteria for unmet need for contraception (capable of pregnancy, sexually active, does not want to become pregnant within the next year, but is currently not using contraception)
* Able to read, write, and speak English
* Willing and able to provide informed consent

Exclusion Criteria:

* Currently pregnant or actively trying to conceive
* Diagnosed infertility (e.g., menopause, tubal ligation, hysterectomy)
* Unable to provide informed consent due to significant cognitive impairment, mental health condition, or substance intoxication
* Unable or unwilling to meet study requirements (e.g., attend sessions, complete assessments)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants who identify as women
Enrollment: 50 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measurement 1: Treatment Completion Rates | Immediately after Session 3 (Week 3)
  Percentage of participants who complete all three intervention sessions, which occur once per week over a three-week period. Completion is defined as attending all sessions and engaging in digital interactive components.
Feasibility Measurement 2: Session Completion Rates | Immediately after each session (Week 1, Week 2, Week 3)
  Percentage of participants who complete each individual session. Completion is defined as attending the full session via videoconference and engaging with digital interactive activities.
Feasibility Measurement 3: Dropout Rates and Reasons for Termination | Immediately after each session (Week 1, Week 2, Week 3)
  Proportion of participants who discontinue participation in the study. Participants who drop out will be asked to complete an exit survey detailing their reasons for withdrawal.
Feasibility Measurement 4: Technical Usability | Immediately after each session (Week 1, Week 2, Week 3)
  Participants will report any technical difficulties they experienced during each session via a brief post-session survey. Measures include ease of use, ability to access materials, and time required to complete digital activities.
Feasibility Measurement 5: Qualitative Feasibility Assessment | 1 week after completion of Session 3 (Week 4)
  Semi-structured qualitative interviews will be conducted to explore participant experiences related to feasibility. Participants will be asked about their ability to complete the intervention, challenges faced, technical usability, and factors influencing session engagement.
Acceptability Measurement 1: Ease of Use | Immediately after each session (Week 1, Week 2, Week 3)
  Participants will rate how easy it was to navigate the intervention, including videoconferencing and digital activities, using a Likert-scale survey (1-5). Mean scores will be calculated across sessions.
Acceptability Measurement 2: Helpfulness | Immediately after each session (Week 1, Week 2, Week 3)
  Participants will assess how useful they found the intervention in supporting behavior change using a Likert-scale survey (1-5). Mean scores will be analyzed for trends across sessions.
Acceptability Measurement 3: Satisfaction | Immediately after each session (Week 1, Week 2, Week 3)
  Overall satisfaction with the intervention will be measured through a Likert-scale survey (1-5), with mean scores reported across sessions.
Acceptability Measurement 4: Qualitative Acceptability Assessment | 1 week after completion of Session 3 (Week 4)
  Semi-structured qualitative interviews will be conducted to explore participant experiences related to acceptability. Participants will be asked about ease of use, perceived helpfulness, satisfaction with the intervention, and suggestions for improvement.
Change from baseline in self-reported primary illicit drug use at 3 months | Baseline and 3-month follow-up
  Participants will report the number of days they used their primary illicit drug (the drug they identify as most problematic) in the past 30 days using the Timeline Followback (TLFB) method. Changes from baseline to 3-month follow-up will be analyzed.
Change from baseline in biologically confirmed illicit drug use at 3 months | Baseline and 3-month follow-up
  Mail-in urine drug tests will be used to verify self-reported illicit drug use. Urine drug test kits will be mailed directly to participants' homes from Phamatech Lab and returned via mail directly to the lab. A positive drug test result will replace a negative self-report. Testing will screen for common substances, including opioids, cocaine, cannabis, and amphetamines.
Change from baseline in the number of participants initiating a contraceptive method highly effective at preventing unintended pregnancy at 3 months | Baseline and 3-month follow-up
  Participants will report whether they have obtained a prescription or started using a contraceptive method considered highly effective at preventing unintended pregnancy, including an implant, intrauterine device (IUD), injection, birth control pill, patch, vaginal ring, or diaphragm. Change from baseline will be assessed.
Change from baseline in effective contraceptive use at 3 months | Baseline and 3-month follow-up
  Participants will report the frequency and consistency of contraceptive use based on manufacturer guidelines. Measures will assess the proportion of sexual acts in which contraception was correctly used over the past 30 days.

SECONDARY OUTCOMES:
Number of participants linked to substance use treatment at 3 months | Baseline and 3-month follow-up
  Linkage to treatment will be measured by the number of participants who report making an appointment for substance use disorder treatment and the number of sessions attended within the three-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa N Slavin, PhD, Principal Investigator — Fairleigh Dickinson University
Locations (1):
- Fairleigh Dickinson University, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data among a vulnerable population, as well as the small sample size (n=50), individual participant data (IPD) will not be shared. Participants are women involved in criminal legal systems with substance use histories, a vulnerable population facing heightened privacy risks. Even with de-identification, there is a concern about the potential for re-identification, particularly given the unique circumstances of participants and the detailed behavioral and health-related data (e.g., drug use) collected. Sharing this data could expose participants to unintended legal, social, or personal consequences. Given these ethical and confidentiality considerations, and in alignment with NIH's guidance on protecting sensitive data, IPD from this study will not be made available for external sharing.